CLINICAL TRIAL: NCT05722405
Title: Exploratory Study of Ixazomib in Combination With Reduced Dose Lenalidomide Versus Ixazomib Alone for Maintenance Treatment of High Risk Multiple Myeloma
Brief Title: Ixazomib Plus Low-dose Lenalidomide Versus Ixazomib Alone for Maintenance Treatment of High Risk Multiple Myeloma
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Affiliated Hospital of Jiaxing University (Other); Huzhou Central Hospital (Other); Lishui Country People's Hospital (Other); Dongyang People's Hospital (Other); Shangyu People's Hospital (Other); Shaoxing People's Hospital (Other); Shaoxing Second Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0215
Record Dates: First submitted 2023-02-01; First posted 2023-02-10 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-11

CONDITIONS: Multiple Myeloma
Keywords: high risk multiple myeloma; Ixazomib; low-dose lenalidomide; maintenance therapy
MeSH Terms: conditions — Multiple Myeloma | interventions — ixazomib; Lenalidomide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ixazomib (Other): Ixazomib as the single drug for maintenance. This group as control arm
  Interventions: Drug: Ixazomib
- Ixazomib plus low-dose lenalidomide (Experimental): Ixazomib combined with low-dose lenalidomide(10mg) for maintenance
  Interventions: Drug: Ixazomib plus low-dose lenalidomide

INTERVENTIONS:
Drug: Ixazomib plus low-dose lenalidomide — Whether Ixazomib combined with low-dose lenalidomide improves the outcome and prognosis of patients with high-risk multiple myeloma as a maintenance treatment option compared to ixazolomib alone
  Other Names: Ninlaro
  Arms: Ixazomib plus low-dose lenalidomide
Drug: Ixazomib — Ixazomib alone
  Other Names: Ninlaro
  Arms: Ixazomib

SUMMARY:
Ixazomib combined with low-dose lenalidomide(10mg) vs Ixazomib alone as maintenance regimen in patients with high-risk multiple myeloma after induction and consolidation of VRD-based regimen.

DETAILED DESCRIPTION:
This study was designed to investigate whether the oral proteasome inhibitor ixazomib combined with low-dose lenalidomide(10mg) as a maintenance regimen could improve the outcome and prognosis of patients with high-risk multiple myeloma after induction and consolidation of VRD-based regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a confirmed diagnosis of symptomatic multiple myeloma with high-risk genetic features (1q21 amplification/t(4;14)/t(14;16)/t(14;20)/17p deletion/TP53 mutation) according to IMWG 2016 criteria.
2. ECOG 0-3
3. After induction and consolidation of the VRD regimen (where patients younger than 65 years of age who are eligible for autologous HSCT and are willing to undergo autologous HSCT collect stem cells and complete autologous HSCT after 3 courses and continue bortezomib or Ixazomib continuous therapy while awaiting transplantation and complete post-transplant consolidation; patients who are not eligible for HSCT regulation or refuse to undergo autologous HSCT go directly to consolidation after induction therapy) and are willing to receive maintenance therapy.
4. Expected survival beyond 6 months
5. Age 18 to 80 years.
6. Adequate renal, hepatic, pulmonary and cardiac function, defined as follows Creatinine clearance (as estimated by Cockcroft-Gault) ≥ 60 ml/min (except for abnormal renal function due to multiple myeloma).

   Serum ALT and AST below 2.5 times the upper limit of normal Total bilirubin below 1.5 times the upper limit of normal Cardiac ejection fraction ≥ 50%, no pericardial effusion confirmed by echocardiography, no clinically significant electrocardiographic findings Absence of clinically significant pleural effusion Baseline oxygen saturation ≥ 95% while indoors
7. Serum or urine pregnancy tests must be negative in women of childbearing potential (women who have undergone sterilization or are at least 2 years post-menopausal may be considered infertile), and patients treated with lenalidomide should have strict contraception and birth control measures.
8. Patients are able to comply with the trial protocol as judged by the investigator.
9. Patients voluntarily participate in this clinical trial, understand the study procedures and are able to sign the informed consent in writing.

Exclusion Criteria:

1. Presence of fungal, bacterial, viral or other infections that are uncontrollable or require IV antimicrobial therapy. Presence of simple urinary tract infection and uncomplicated bacterial pharyngitis, after consultation with the investigator, if responsive to active treatment.
2. Known presence of HIV or a history of hepatitis B (HBsAg positive) or viral hepatitis C (anti-HCV positive) infection. A history of treated hepatitis B or hepatitis C is allowed if a viral load undetectable by quantitative PCR and/or nucleic acid testing is present.
3. A history of thrombosis within six months.
4. presence of a history of malignancy other than carcinoma in situ (e.g., cervical, bladder, breast, thyroid), except in patients who have not had an episode for at least 3 years
5. Patients with uncontrolled arrhythmias and a history of myocardial infarction, cardiac angioplasty or stenting, unstable angina or other clinically significant cardiac disease within 12 months of enrollment.
6. The presence of a significant immunodeficiency.
7. The presence of any medical condition that may interfere with the assessment of the safety or efficacy of the investigational treatment.
8. A history of severe hypersensitivity reactions to this investigational drug.
9. Any pregnant or breastfeeding female of childbearing potential.
10. Male and female subjects who are unwilling to use birth control within 6 months from the time of signing the consent form until the completion of the administration of this study.
11. Subjects who, in the judgment of the investigator, are unlikely to complete all study visits or procedures required by the protocol, including follow-up visits or compliance with the requirements for participation in the study.
12. History of autoimmune disease (e.g., Crohn's disease, rheumatoid arthritis, systemic lupus erythematosus) within the past 2 years that causes end-organ damage or requires systemic immunosuppressive/systemic disease-modifying drugs.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | through study completion, a average of 1 year
  PFS is defined as the time from the date of first dose of study drug to the first occurrence of PD as evaluated by the investigator or death from any cause, whichever occurs first. PD is defined as >=25% increase from lowest value in serum M component or urine M-component; difference between involved and uninvolved free light chain (FLC) levels (absolute increase >10 mg/dL); bone marrow plasma cell percent >/=10%; new bone lesions or soft tissue plasmacytomas development or definite increase in existing bone lesions/soft tissue plasmacytomas size; hypercalcaemia development.

SECONDARY OUTCOMES:
Very Good Partial Response (VGPR) + Complete Response (CR) Rate | through study completion, a average of 1 year
  Using IMWG criteria
Overall Survival (OS) | through study completion, a average of 1 year
  OS is measured as the time from the date of first dose of study drug to the date of death.
Percentage of Participants with Adverse Events (AEs) | through study completion, a average of 1 year
  Adverse events are defined as any unfavorable and unintended sign, symptom or disease temporally associated with the use of a medicinal product reported from first dose of study drug through 30 days after the last dose of study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Yang Xu, Dr., Study Director — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- Yang Xu, Hangzhou, Zhejiang, China